CLINICAL TRIAL: NCT06127589
Title: An Integrated Smoking Cessation Intervention Model of Brief Advice, Nicotine Replacement Therapy and Mobile Health Support for Smoking Parents to Increase Abstinence and Protect Children from Tobacco Smoke Exposure: a Randomized Controlled Trial
Brief Title: The "Quit-for-Kids" Project: to Increase Abstinence and Protect Children from Tobacco Smoke Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QFK
Record Dates: First submitted 2023-10-10; First posted 2023-11-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation; Second Hand Tobacco Smoke
Keywords: Smoking Cessation; Second Hand Smoke Exposure; Children Health; Mobile Health Intervention; Nicotine Replacement Therapy; Family-based Intervention
MeSH Terms: conditions — Smoking Cessation | interventions — Crisis Intervention; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief cessation advice + Nicotine replacement Therapy + Instant Messaging + Financial Incentives (Experimental): Participants will receive a special designed evidence-based intervention using health advice, behavioral and pharmacological support, mobile health technologies, and awareness building (highlight harms) based on the biofeedback results of SHS exposure in the child. A selected sample of 50 families will receive environmental assessment-derived intervention, including results interpretation and health advice, which will be provided via phone calls for the 50 families within 1 week after the data collection.
  Interventions: Behavioral: Brief cessation advice (AWARD); Drug: Nicotine Replacement Therapy (NRT); Behavioral: Instant messaging Support (IM); Behavioral: Financial Incentive (FI); Behavioral: Self-help smoking cessation booklet; Behavioral: Environmental assessment derived intervention
- Brief cessation advice (AWARD) + Waitlist for same intervention (Active Comparator): Participants in the control group will receive the same AWARD brief advice model, self-help booklet at baseline, and financial incentives for validated abstinence at 3- and 6-month follow-up. After the 6-month follow-up, participants who continued to smoke will receive the remaining intervention components: 1-week sampling of NRT and 3 months instant messaging chat-based personalized psychosocial and behavioural counselling for quitting. Participants who validated abstinence at the 12 months or actively engaged in mobile Health counselling will also receive the financial incentives of HK$ 500 and HK$ 200, respectively (waitlist control).
  Similar to the Intervention group, environmental assessment derived intervention, including results interpretation and health advice, will be provided via phone calls for the 50 families within 1 week after the data collection.
  Interventions: Behavioral: Brief cessation advice (AWARD); Behavioral: Self-help smoking cessation booklet; Behavioral: Environmental assessment derived intervention

INTERVENTIONS:
Behavioral: Brief cessation advice (AWARD) — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refuse to set a quit date).
  Other Names: Brief Advice (BA)
Drug: Nicotine Replacement Therapy (NRT) — 1-week sampling of Nicotine Replacement Therapy (NRT) will be provided to support quit attempt. Full pharmacological treatment (12-week) will be available if needed.
  Other Names: NRT
  Arms: Brief cessation advice + Nicotine replacement Therapy + Instant Messaging + Financial Incentives
Behavioral: Instant messaging Support (IM) — Chat-based mHealth personalized psychosocial and behavioural counselling (smoking cessation and SHS exposure reduction messages will be derived from previously tested interventional studies) using baseline children health and biofeedback data to support quitting throughout the intervention period of 3 months.
  Other Names: IM
  Arms: Brief cessation advice + Nicotine replacement Therapy + Instant Messaging + Financial Incentives
Behavioral: Financial Incentive (FI) — A financial incentive (vouchers) of HK$ 500 will be provided for biochemically validated smoking abstinence at 3- and 6-month follow-up. Considering a possibly low engagement rate of the smokers in mHealth-based support (17% in our previous trial, non-engagement mostly due to busy work), additional HK$ 200 will be provided for participants who actively engaged in the mHealth counselling (defined by have discussed quitting process for >2 times) at 3-month follow-up.
  Other Names: FI
  Arms: Brief cessation advice + Nicotine replacement Therapy + Instant Messaging + Financial Incentives
Behavioral: Self-help smoking cessation booklet — A well-designed self-help booklet will be provided to guide and provide detailed information on smoking cessation. The contents include information about the benefits of quitting, smoking and diseases, methods to quit, how to handle withdrawal symptoms, declaration of quitting, etc.
  Other Names: Self-help material
Behavioral: Environmental assessment derived intervention — In a selected subgroup of 50 families with an additional signed consents, four home visits will be done to: 1. Setup an indoor air quality (IAQ) monitor to collect 24hr air quality data (2 weeks), 2. Collect the monitor for data retrieval, 3. Setup the monitor at 6 months follow-up (2 weeks), 4. Collect the monitor for data retrieval.
  Environmental assessment derived intervention, including results interpretation and health advice, will be provided via phone calls for the 50 families within 1 week after the data collection.

SUMMARY:
This project aims to test the effectiveness of an integrated intervention of brief cessation advice (AWARD), Nicotine Replacement Therapy, and Instant Messaging support compared with waitlist control participants among adult daily smokers who lived with their children and non-smoking partners.

DETAILED DESCRIPTION:
Background: Around 40% of children worldwide were exposed to secondhand smoke (SHS). Despite reaching a single-digit smoking prevalence of 9.5% in 2022, about one in three children in Hong Kong (36.2%) are still exposed to SHS, mostly at home. Especially children from deprived households, suffer from a higher risk of more pervasive SHS exposure. Aim: The project aims to apply evidence-based interventions to increase smoking cessation and reduce SHS exposure in children of disadvantaged families. The specific objectives of the study are (1) to evaluate the effectiveness of a novel, family-based intervention model in increasing smoking cessation and reducing SHS exposure in children of disadvantaged families, (2) to alert parents in recognizing their child's exposure level and take actions in protecting their child from exposure, (3) to advocate for the adoption of this resource-efficient intervention model in Non-Governmental Organizations(NGOs), District Health Centre Express(DHC/Es), and other smoking cessation service providers in Hong Kong.

Methods: A family-based smoking cessation that collect comprehensive biochemical and environmental data of SHS exposure, and apply evidence-based interventions to prevent the SHS exposure and support quitting in deprived households. Two domains of outcome will be assessed: (1) Effectiveness and overall impact of smoking cessation intervention. (2) Cost-effectiveness analysis and qualitative interviews to estimate the scalability and mechanisms of interventions.

Procedure: Participants will be actively recruited through different channels including direct referral from Non-Governmental Organizations (NGOs) with social housing schemes, referral and recruitment from District Health Centre (DHC), community-based recruitment activities in smoking hotspots, and online advertisement on search engines and social media sites. The eligibility of smokers and non-smokers will be assessed by counselors and invited to join the randomized controlled trial and allocated to one of the groups of the smoking cessation intervention. 6 follow ups at 1 week, 1,2,3,6,12 months will be conducted to both smokers and non-smokers to reveal their SHS exposure level and smoker's quitting progress.

Hypothesis: We hypothesize that the assessment-guided intervention will lead to significant increases in rates of smoking cessation in the intervention group than the control group. Another hypothesis to be investigated is that designated intervention messages are effective to reduce the level of SHS participants and their family members exposed to.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 tobacco stick (includes HTP) per day or use e-cigarette daily in the preceding 3-month and verified by exhaled carbon monoxide level of 4ppm (parts per million) or above, assessed by a validated Carbon monoxide Smokerlyzer®
* Living with at least one child of primary 6 or below (aged 12 or below)
* Living with at least one non-smoking family member
* Living in deprived households (monthly household income of less than the median of household monthly income in Hong Kong, HK$ 28,000, or living in subdivided flats or social housing)
* Able to communicate in Chinese (including reading Chinese in IM)
* Able to use the instant messaging tool (e.g., WhatsApp, WeChat) for communication

Exclusion Criteria:

* Those who have communication barriers (either physically or cognitively)
* Those who are currently participating in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated abstinence | 6-month after recruitment
  Defined as exhaled carbon monoxide level <4ppm and saliva cotinine level ≤30ng/ml

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate (for smokers) | 3- and 6-month after recruitment
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported reduction rate (for smokers) | 3- and 6-month after recruitment
  Defined by at least 50% reduction in baseline daily number of cigarettes.
Self-reported intention to quit (for smokers) | 3- and 6-month after recruitment
  Defined by readiness to quit in 30 days.
Smoking cessation service use (for smokers) | 3- and 6-month after recruitment
  The number of calling a hotline of the smoking cessation services, booking an appointment, smoking cessation clinic attendance, and counseling session attendance.
Self-rated health (for smokers) | 3- and 6-month after recruitment
  Self-reported health status will be measured using a single-item scale (in general, would you say that your health is excellent, very good, good, fair, or poor?")
Children's secondhand smoke exposure (for children) | 3- and 6-month after recruitment
  The children's SHS exposure will be assessed by the nicotine or cotinine level in urine, saliva, or hair using isotope dilution liquid chromatography and tandem mass spectrometry with a limit of detection of < 50 parts per trillion.
Academic performance (for children) | 3- and 6-month after recruitment
  Participant's academic performance will be assessed by "In general, would you say your academic performance is Excellent/Very good/Good/Fair/Poor?"
Cognitive function (for children) | 3- and 6-month after recruitment
  Participant's cognitive function will be assessed by "In general, would you say your cognitive function is Excellent/Very good/Good/Fair/Poor?"
Self-reported secondhand smoke exposure (for children and family member) | 3- and 6-month after recruitment
  Self-reported secondhand smoke exposure will be measured using a single-item scale (In the past week, have you inhaled secondhand smoke in your home? No or Yes, for___days)
Quality of life (for smokers and family member) | 3- and 6-month after recruitment
  Quality of life will be measured by Health-related Quality of life-short form (SF12), which contains eight dimensions (General Health, Physical Function, Role Physical, Bodily Pain, Vitality, Social Functioning, Role Emotional, and Mental Health). The scale ranges from 0 to 100, with the higher the score, the better and healthier they feel subjectively.
Depression and anxiety (for smokers, family member and children) | 3- and 6-month after recruitment
  The Patient Health Questionnaire-4 (PHQ-4) will be used to measure depression and anxiety. The 4-item questionnaire consists of a 2-item depression sub-scale and 2-item anxiety sub-scale. The questions are answered on a four-point Likert Scale. The sum of the scores is categorized into normal (0-2), mild (3-5), moderate (6-8) and severe (9-12). The total score of 3 or greater on each sub-scale suggest depression or anxiety, respectively.
Family well-being (for smokers, family member and children) | 3- and 6-month after recruitment
  Family well-being will be measured by family health, harmony, and happiness (3Hs): three separate questions asked, "How healthy/harmonious/happy do you think your family is?" and will be answered using an 11-point scale ranging from 0 to 10, with higher scores indicating higher level of family well-being.
Respiratory symptoms (for smokers, family member and children) | 3- and 6-month after recruitment
  Respiratory symptoms will be measured by a single-item scale (In the past week, if you have had any of the following symptoms, with the response of having trouble with your eyes, sore throat, cough, shortness of breath, runny nose, loss of appetite, and rapid heartbeat).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China